CLINICAL TRIAL: NCT01503554
Title: Multidisciplinary Care Transition Intervention - Cardinal Health Grant
Brief Title: Combined Social Worker and Pharmacist Transitional Care Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Shannon Sims, MD, MD, PhD, Rush University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11010702-IRB01; Care Trans-IT (Other Grant/Funding Number: Cardinal Health)
Record Dates: First submitted 2011-12-30; First posted 2012-01-04 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Patient Admission; Patient Discharge
MeSH Terms: interventions — 2-ethylidene-1,5-dimethyl-3,3-diphenylpyrrolidine; Pharmacists; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Worker + Pharmacist Intervention (Experimental): Intervention arm offering enhanced services from a social worker and a pharmacist post-discharge
  Interventions: Behavioral: Combined Social Worker and Pharmacist Program
- Usual Care (Experimental): Patients receiving usual care will have a medication reconciliation performed by a physician or nurse during their hospital stay. No further support or interventions are provided post discharge.
  Interventions: Behavioral: No Intervention: Usual Care

INTERVENTIONS:
Behavioral: Combined Social Worker and Pharmacist Program — Physician or nurse performs a med rec during hospital stay Clinical pharmacist completes an additional med rec of home meds, assesses med-related risks, and provides education After discharge, a Master's prepared social worker contacts the patient and conducts an assessment from a psychosocial perspective to identify any unmet needs.
  Pharmacist will be available to patients should they have any medication-related questions post-discharge
  Other Names: EDPP Plus Pharmacist
  Arms: Social Worker + Pharmacist Intervention
Behavioral: No Intervention: Usual Care — Patient receives usual care upon discharge from the hospital.
  Other Names: Control Group
  Arms: Usual Care

SUMMARY:
In an effort to improve care coordination and reduce hospital readmissions, Rush University Medical Center developed the Combined Social Worker and Pharmacist Program, which targets both the psychosocial and clinical risk factors that can lead to rehospitalization. This study will evaluate the impact of this program on 30-day same hospital readmission rates and total cost of care.

DETAILED DESCRIPTION:
If a patient is enrolled in the Combined Social Worker and Pharmacist Program their care will differ from usual care in a number of different ways. First, while the patient is in the hospital, an interdisciplinary group of providers will round on the patient on a regular basis. This interdisciplinary team will be composed of an attending physician, clinical pharmacist, nurse, case manager, and social worker, who will all evaluate the patient's needs from a variety of perspectives to ensure that the patient is prepared for discharge and self-manage post-discharge. During the patient's hospital stay, a clinical pharmacist will also conduct a detailed medication reconciliation of home medications, assess medication-related risks, and provide relevant education to patients participating in the program. After the patient is discharged from Rush University Medical Center, a Master's prepared social worker will then contact the patient and conduct an assessment from a psychosocial perspective to identify any unmet needs. Lastly, a clinical pharmacist will be available to patients enrolled in the Combined Social Worker and Pharmacist Program, should they have any medication-related questions post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Planned discharge to home or home health
* English-speaking
* At least one of the following risk factors:
* Use of high risk medication(s): Anti-coagulant therapy, dual ASA/plavix therapy, anticholinergic agent, digoxin, opioids, psychotropic medications, or erythrocyte stimulating factor
* Clinical risk factor: Depression, fall risk, limited functional capacity, substance abuse, dementia
* Psycho-social risk factor: high care giver burden, family conflict, limited health literacy, lives alone, significant patient stress, transportation concerns, health care scheduling concerns, inadequate emotional support.

Exclusion Criteria:

* Hospice
* Solid organ transplant
* End-stage renal disease
* Current chemotherapy or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
30-day Same Hospital Readmission Rate | 30 days following hospital discharge

SECONDARY OUTCOMES:
Total Cost of Care | 30 days following hospital discharge
  Outcome measure seeks to capture the total cost of care within 30 days of discharge (i.e., costs associated with hospital readmissions, ED visits, outpatient visits, and program costs, if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Sims, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States